CLINICAL TRIAL: NCT04436458
Title: Phase 2, Multicentre, Randomized, Double Blind, 2 Arms Placebo-controlled Study in Adults With Moderate COVID-19 With Gastrointestinal Signs and Symptoms
Brief Title: Niclosamide In Moderate COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor asset acquired by another pharma company who opened their own IND for this compound. First Wave Bio never started this study in the US or ex-US.
Sponsor: Entero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FW-COV-002
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-02

CONDITIONS: COVID
MeSH Terms: interventions — Niclosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Niclosamide (Experimental): Continued SOC therapy together with Niclosamide tablets for 14 days
  Interventions: Drug: Niclosamide Oral Tablet
- Placebo (Placebo Comparator): Continued SOC therapy together with placebo tablets matching niclosamide
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niclosamide Oral Tablet — Continued SOC therapy together with niclosamide TID for 14 days
  Arms: Niclosamide
Drug: Placebo — Continued SOC therapy together with placebo tablets matching niclosamide for 14 days
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicentre, randomized, double blind, 2 arm placebo-controlled study in adults with moderate COVID-19 with gastrointestinal signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for treatment of COVID-19 with or without pneumonia, who are expected to remain in hospital at least seven days after the randomization and who accept continuing to be assessed for the study procedures (home or outpatient unit) up to 6 weeks in case of discharge.
* Patients who prior to developing COVID-19 usually have normal bowel habits defined as at least 3 stools per week and no more than 3 stools per day.
* SARS-CoV-2 infection confirmed by RT-PCR in rectal swab (or stool test) ≤2 days before randomization by local or central lab.
* Diarrhea defined as at least 3 watery stools in the last 24 hours prior to enrolment

Exclusion Criteria:

* At the time of randomization patients requiring ICU admission or patients with severe respiratory insufficiency requiring mechanical ventilation or with rapid worsening of respiratory function leading to expectation for mechanical ventilation or ICU admission.
* Evidence of rapid clinical deterioration or existence of any life-threatening co-morbidity or any other medical condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the rate of faecal SARS-CoV-2 virus clearance (rectal swab or stool sample) assessed by RT-PCR in the niclosamide group, compared to the placebo group | From Day 1 to 42